CLINICAL TRIAL: NCT06147700
Title: Identifying Molecular Determinants of Infertility in Men (MODIFY)
Status: Completed | Type: Observational
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Principal Investigator, Candida Vaz, Principal Investigator, Senior research scientist, Institute for Human Development and Potential (IHDP), Singapore
Other Study IDs: 2023-085
Record Dates: First submitted 2023-09-25; First posted 2023-11-28 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy fertile male: No intervention for this study.
- Healthy infertile male: No intervention for this study.

SUMMARY:
The purpose of this study is to understand the underlying mechanisms of infertility caused by unknown factors. The investigator propose to identify small non-coding RNA (sncRNA) biomarkers of infertility and advance towards developing a more accurate and robust approach for infertility diagnosis.

DETAILED DESCRIPTION:
The goal of the study is to identify small non-coding RNA signatures of infertility in men through the comparison of sperm sncRNA profiles from around 100 men (21-50 years of age). The participants will be classified into fertile and infertile groups by the conventional method.

Through the project, the investigator intends to understand the underlying mechanisms of idiopathic infertility. By utilizing semen as liquid biopsy, through sperm sncRNA profiling and comparison (infertile vs fertile). The investigator proposes to identify the sncRNA (miRNAs, piRNAs and tRFs) as biomarkers of infertility.

The investigator proposes to generate a validated signature of sncRNAs that will help in selecting high quality sperms for IVF.

ELIGIBILITY:
Inclusion Criteria

* Male, aged 21 - 50 years old
* Proficient in English language
* Willing to comply to study protocol
* Able to provide written informed consent

Exclusion Criteria

* Current and/or previous diagnosis of Tuberculosis, Acquired immunodeficiency syndrome (AIDs), and other sexually transmitted diseases
* Experiencing severely limited mobility (eg. Wheelchair bound, need walking aid)
* Diagnosed with severe unstable mental conditions (eg. Dementia, or cognitive impairment)
* Alcohol or drug abuse

Ages: 21 Years to 50 Years | Sex: Male
Age Groups: Adult
Gender Based: Yes — Healthy males
Study Population: Healthy male in the general population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Semen/Sperm quantity analysis | 1 week
  sperm count and concentration
Semen/Sperm quality analysis | 1 week
  semen pH, semen volume, sperm motility, sperm morphology, sperm vitality
Fertility classification | 1 week
  Classification into fertile/infertile groups based on the fertility measures.
Sperm RNA extraction and sequencing | 3 months
  Sperm RNA extraction and sequencing

SECONDARY OUTCOMES:
Expression profiling of sncRNA | 3-6 months
  Counts of miRNA, piRNA, tRF from the sequenced data through Bioinformatics analysis. All three sncRNA will be quantified from the RNA sequencing data using bioinformatics tools, with the same unit of measure.
Comparison of the expression profiles | 3-6 months
  Comparison of the expression profiles between the two groups (infertile vs fertile)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Development Research Centre (HDRC), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
PDPA law in Singapore

REFERENCES:
- [Background] Soubry A. POHaD: why we should study future fathers. Environ Epigenet. 2018 Apr 26;4(2):dvy007. doi: 10.1093/eep/dvy007. eCollection 2018 Apr. PMID 29732171
- [Background] Donkin I, Barres R. Sperm epigenetics and influence of environmental factors. Mol Metab. 2018 Aug;14:1-11. doi: 10.1016/j.molmet.2018.02.006. Epub 2018 Feb 27. PMID 29525406
- [Background] Khatun A, Rahman MS, Pang MG. Clinical assessment of the male fertility. Obstet Gynecol Sci. 2018 Mar;61(2):179-191. doi: 10.5468/ogs.2018.61.2.179. Epub 2018 Mar 5. PMID 29564308
- [Background] Cao XW, Lin K, Li CY, Yuan CW. [A review of WHO Laboratory Manual for the Examination and Processing of Human Semen (5th edition)]. Zhonghua Nan Ke Xue. 2011 Dec;17(12):1059-63. Chinese. PMID 22235670
- [Background] Zhang Y, Shi J, Rassoulzadegan M, Tuorto F, Chen Q. Sperm RNA code programmes the metabolic health of offspring. Nat Rev Endocrinol. 2019 Aug;15(8):489-498. doi: 10.1038/s41574-019-0226-2. Epub 2019 Jun 24. PMID 31235802
- [Background] Vashisht A, Gahlay GK. Using miRNAs as diagnostic biomarkers for male infertility: opportunities and challenges. Mol Hum Reprod. 2020 Apr 24;26(4):199-214. doi: 10.1093/molehr/gaaa016. PMID 32084276
- [Background] Alves MBR, Celeghini ECC, Belleannee C. From Sperm Motility to Sperm-Borne microRNA Signatures: New Approaches to Predict Male Fertility Potential. Front Cell Dev Biol. 2020 Aug 21;8:791. doi: 10.3389/fcell.2020.00791. eCollection 2020. PMID 32974342
- [Background] Abu-Halima M, Hammadeh M, Backes C, Fischer U, Leidinger P, Lubbad AM, Keller A, Meese E. Panel of five microRNAs as potential biomarkers for the diagnosis and assessment of male infertility. Fertil Steril. 2014 Oct;102(4):989-997.e1. doi: 10.1016/j.fertnstert.2014.07.001. Epub 2014 Aug 6. PMID 25108464
- [Background] Cui L, Fang L, Shi B, Qiu S, Ye Y. Spermatozoa micro ribonucleic acid-34c level is correlated with intracytoplasmic sperm injection outcomes. Fertil Steril. 2015 Aug;104(2):312-7.e1. doi: 10.1016/j.fertnstert.2015.05.003. Epub 2015 Jun 6. PMID 26051092
- [Background] Hua M, Liu W, Chen Y, Zhang F, Xu B, Liu S, Chen G, Shi H, Wu L. Identification of small non-coding RNAs as sperm quality biomarkers for in vitro fertilization. Cell Discov. 2019 Apr 9;5:20. doi: 10.1038/s41421-019-0087-9. eCollection 2019. No abstract available. PMID 30992999

DOCUMENTS (1):
  • Informed Consent Form (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT06147700/ICF_000.pdf